CLINICAL TRIAL: NCT03937297
Title: A Culturally Appropriate Multimodal Non-pharmacological Intervention for Chinese People With Mild-to-Moderate Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Alzheimer's Disease Association (Unknown); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17612418
Record Dates: First submitted 2019-04-16; First posted 2019-05-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Dementia
Keywords: non-pharmacological; intervention; culturally appropriate; Chinese; cognitive stimulation therapy; Six Arts; dementia; CST
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor would not be told if the participant is in the intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Six Arts intervention
  Interventions: Behavioral: Six Arts
- Arm 2 (Experimental): Cognitive Stimulation Therapy (CST)
  Interventions: Behavioral: Cognitive Stimulation Therapy (CST)
- Arm 3 (Active Comparator): Usual care (control group)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Six Arts — The Six Arts intervention is a 24 session, twice a week intervention protocol. There will be four sessions per "Art", with specific sequence designed to enhance group dynamic and create harmony. Each session starts with a 15 minutes warm-up exercise, followed by the Six Art theme activity. The program design emphasizes on integrated cognitive, physical, and social activities covering all domains of Six Arts.
  Arms: Arm 1
Behavioral: Cognitive Stimulation Therapy (CST) — The CST to be used involve 24 sessions of theme activities, twice a weekly intervention protocol. It is modified into CST-Hong Kong for activities that are not applicable in Hong Kong Chinese culture (e.g. word games involving alphabets)
  Arms: Arm 2
Behavioral: Usual Care — usual dementia care provided by participating center
  Arms: Arm 3

SUMMARY:
This is a mixed-methods research that includes a single-blind three-arms randomized control trials and a focus group study. The quantitative study aims to investigate the additional clinical benefits of the Six Arts intervention over an evidence-based non-pharmacological intervention translated from western culture, cognitive stimulation therapy (CST). The qualitative part aims to explore the acceptance and understanding of family caregiver of the Six Arts intervention and CST.

It is hypothesized that 1) the group who have received Six Arts intervention would show superior quality of life; 2) both Six Arts and CST groups would show superior cognitive improvement compared with usual care; 3) the Six Arts group would show greater improvement in behavioral and neuropsychological symptoms and functioning compared with the groups receiving CST or usual care.

DETAILED DESCRIPTION:
Dementia is a disabling chronic condition affecting over 47 million people worldwide. Chinese population will be one of the main driver in the increasing trend in dementia prevalence. Accumulating evidence suggests effectiveness of certain non-drug interventions in maintaining cognition and quality of life in people with mild-to-moderate dementia, such as cognitive stimulation therapy (CST). These interventions are designed and tested in western populations with issues of cultural adaptation when applied in Chinese. Culturally appropriate and effective interventions for Chinese people with mild-to-moderate dementia are lacking.

The Six Arts stem from ancient Confucian philosophy, which promotes behaviours that can impact on multiple mind-body functional domains. These domains correspond to social, physical, and cognitive activities with theoretical basis and empirical evidence of benefits in cognition, functioning, and quality of life. Using the Six Arts as a cultural framework, a group-based multimodal intervention has been developed in Hong Kong for Chinese people with mild-to-moderate dementia.

The study will recruit 240 people with mild-to-moderate dementia in a randomized single-blind controlled trial consisting of three groups: (1) Six Arts intervention; (2) CST; and (3) usual care. Neuropsychological and clinical assessments will be conducted at randomization (T0/baseline) and upon completion of the 24-session, twice-weekly intervention (T1/3 months), by an assessor unaware of group membership. Focus groups will be conducted after completion of the intervention in 60 family caregivers who have observed at least one session of the Six Arts intervention or CST.

This study will provide evidence on the effectiveness of two intervention protocols with potentials for large-scale implementation in the growing Chinese population with dementia.

ELIGIBILITY:
People with dementia:

Inclusion Criteria:

* aged 60 or above
* have clinical diagnosis of dementia or a Clinical Dementia Rating (CDR) of 1-2 suggestive of mild-to-moderate disease;
* able to communicate and understand communication, see and hear well enough to participate in a meaningful assessment;
* person with dementia and/or his/her caregiver can provide informed consent

Exclusion Criteria:

* suffering from major physical illness or disability that affect participation;
* had experience with the 24-session of CST or Six Arts intervention protocols

Caregivers (for the focus group study)

Inclusion Criteria:

* provide care to the person of dementia for more than 8 hours per week
* have observed at least one intervention session of either CST or Six Arts intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life of people with dementia | T0 (baseline), T1 (up to 4 months)
  measure by using a 13-item self-rating and proxy rating scale, the Quality of Life in Alzheimer's Disease (QoL-AD)
Changes in cognitive performance | T0 (baseline), T1 (up to 4 months)
  measure by using the Alzheimer's Disease Assessment Scale - Cognitive section (ADAS-Cog), a standard cognitive test commonly used in clinical trials for people with dementia

SECONDARY OUTCOMES:
CDAD | T0 (baseline), T1 (up to 4 months)
  measure the changes in functioning by using the Chinese version of the Disability Assessment for Dementia (CDAD), a 11-item scale that evaluates the basic and instrumental activities in daily activities of elderly people with dementia
NPI-Q | T0 (baseline), T1 (up to 4 months)
  measure the changes in behavioral and psychological symptoms of dementia by using the Neuropsychological Inventory Questionnaire (NPI-Q), a 12-item informant-based interview

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Yan, Gloria Wong, PhD, Principal Investigator — non-med affiliation
Locations (1):
- The University of Hong Kong, Hong Kong, Non-US Or Canadian Address, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Not planning to share the data